CLINICAL TRIAL: NCT04137068
Title: Sedentary Behavior, Cardiovascular Function, and Sleep
Acronym: PACE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Oregon Health and Science University (Other)
Responsible Party: Principal Investigator, Saurabh Thosar, Principal Investigator, Oregon Health and Science University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: STUDY00020458
Record Dates: First submitted 2019-10-15; First posted 2019-10-23 (Actual); Last update posted 2022-08-05 (Actual); Status verified 2022-08

CONDITIONS: Sedentary Behavior; Cardiovascular Function; Sleep
Keywords: Physical Activity; Sleep; Sedentary; Cardiovascular
MeSH Terms: conditions — Sedentary Behavior; Motor Activity

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Sedentary to Active (Other): Participants will visit the research laboratory for baseline measurements at visit 1 after wearing a pedometer for one week and maintaining their typical level of physical activity. After the baseline visit, participants will reduce their step count by more than half for two weeks. Participants will visit the laboratory once every week during the 2 week interventional period for a total of 3 visits.
  Interventions: Behavioral: Reduced Activity

INTERVENTIONS:
Behavioral: Reduced Activity — Participants reduce their activity level to <5,000 steps/day and <50 % of baseline steps.
  Other Names: Sedentary Behavior

SUMMARY:
This is an interventional study that will examine how sedentary behavior (decreased physical inactivity) over time affects cardiovascular health (i.e. heart rate and blood pressure) and sleep quality/duration.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

1. To test the hypothesis that two weeks of sedentary behavior will progressively impair vascular endothelial function.

2: To test the hypothesis that increasing sedentary behavior will decrease total sleep duration and sleep efficiency.

3: To test the hypothesis that two-weeks of sedentary behavior will progressively increase 24-h blood pressure and reduce nocturnal blood pressure dipping.

OUTLINE:

After a baseline period, participants will become more inactive and also come in for 4-h uninterrupted sitting visits. Cardiovascular, activity, and sleep measures will be taken throughout.

ELIGIBILITY:
Inclusion Criteria:

* Ages 20-80y
* Lean and overweight (BMI 18.5-40 kg/m2)
* No acute, chronic, or debilitating medical conditions
* No prescription/non-prescription medications or drugs of abuse
* Limited weight training or intense exercise (swimming, CrossFit)
* Non-smoker
* Average level of daily physical activity (8,000-12,499 steps/day)
* Persons who fit all the above criteria and are suitable based on a medical history and health habits questionnaire, sleep profiling questionnaire, and electrocardiogram and clinical biochemical screening tests of blood and urine may be eligible to participate.

Exclusion Criteria:

* Persons with any acute, chronic, or debilitating medical condition except pre-hypertension and/or mild to moderate sleep apnea will be excluded.
* Persons with any symptoms of acute or active illness (e.g. fever, leukocytosis) will be excluded.
* Persons with a history of severe psychiatric illness or psychiatric disorders will be excluded.
* Persons with a history of regular night/or rotating shift work, or who have traveled more than three time zones during the one month prior to the study will be excluded.
* Pregnant persons, decisionally impaired adults, and prisoners will be excluded.

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2019-11-13 (Actual); Primary Completion 2023-03-31 (Estimated); Study Completion 2023-03-31 (Estimated)

PRIMARY OUTCOMES:
Endothelial Function | 3 weeks
  Investigators will measure endothelial function as flow-mediated dilation at baseline, and each hour of the 3-hour sitting trials.
Oxidative stress | 3 weeks
  Oxidative stress will be measured using malondialdehyde adducts (MDA) from Ethylenediaminetetraacetic acid (EDTA) plasma.
Endothelin-1 | 3 weeks
  Endothelin 1 (ET-1) will be measured from Ethylenediaminetetraacetic acid (EDTA) plasma.
Heart rate | 3 weeks
  During the weekly trials, heart rate will be measured as beats per minute while participants are in a seated position during the prolonged sitting period.
Blood pressure | 3 weeks
  During the weekly trials, blood pressure will be measured as systolic over diastolic in a seated position in the dominant arm
24-hour BP measurement | 3 weeks
  Investigators will measure 24-hour ambulatory blood pressure monitoring (AMBP, Spacelabs, Inc) at baseline and for 24-h before each in-lab visit.
Sleep duration | 3 weeks
  Sleep duration will be scored from the ActiGraph and correlated with the sleep and activity diary.
Sleep efficiency | 3 weeks
  Sleep efficiency will be scored from the ActiGraph and correlated with the sleep and activity diary.
Activity | 3 weeks
  Activity will be scored from the ActiGraph and correlated with the sleep and activity diary.
Activity Perception | 3 weeks
  Activity perception will be measured before each prolonged sitting trial using an Activity Perception questionnaire (Perception of Current Activity Questionnaire). The questionnaire has 7 questions with answers ranging from 1 to 5. The range of scores is from 7 to 35, with 7 suggesting a strong negative perception of current activity, and 35 suggesting a strong positive perception of current activity.

CONTACTS AND LOCATIONS:
Overall Officials: Saurabh Thosar, Dr., Principal Investigator — Oregon Institute of Occupational Health Sciences
Locations (1):
- Oregon Institute of Occupational Health Sciences, Portland, Oregon, United States

IPD SHARING:
Plan to Share IPD: No